CLINICAL TRIAL: NCT00618969
Title: A Phase II Study of Peripheral Blood Stem Cell Transplantation (PBSCT)From Haploidentical Related Donors for Treatment of Hematologic Malignancies and Hematopoietic Failure States
Brief Title: Peripheral Blood Stem Cell Transplantation (PBSCT)From Haploidentical Related Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO 07-122; NCT00840424 (obsolete NCT alias)
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Hematologic Neoplasms; Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Multiple Myeloma
Keywords: Haploidentical; peripheral blood stem cell transplantation; leukemia; myeloma; Hodgkin's disease; non-Hodgkin's lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Multiple Myeloma; Leukemia; Neoplasms, Plasma Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Busulfan; Melphalan; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical allogeneic PBSC transp (Experimental): Non-myeloablative preparative regimen (reduced-intensity) of busulfan, melphalan and alemtuzumab followed by a haploidentical-related peripheral blood stem cell transplant.
  Interventions: Other: haploidentical allogeneic PBSC transp

INTERVENTIONS:
Other: haploidentical allogeneic PBSC transp — Days -5 and -4: IV busulfan 3.2 mg/kg/dose daily for 2 days
  Day -3: IV melphalan 100 mg/m2 as a single dose
  Days -2 and -1: IV alemtuzumab 30 mg/dose daily for 2 days
  Day 0: Transplantation of haploidentical related allogeneic peripheral blood stem cells (PBSCs)- target cell dose 10 x 106 donor CD34+ cells per kilogram of recipient weight
  Other Names: Myleran,; Busulfex,; Busulphan; Alkeran,; L-PAM, L-Sarcolysin,; Phenylalanine Mustard; MABCAMPATH®,; CAMPATH®; partially matched family related donor transplant

SUMMARY:
The purpose of this study is to transplant haploidentical related peripheral blood stem cells (PBSCs) that come from a relative such as a parent, sibling, a child or other relative who has a half-matched tissue type with the recipient (rather than being completely matched) following administration of a reduced-intensity regimen of busulfan, melphalan and alemtuzumab.

DETAILED DESCRIPTION:
Fewer than 35% of patients who might benefit from allogeneic HCT have an HLA-identical sib. Transplantation of peripheral blood stem cells (PBSCs) or bone marrow (BM)from HLA-matched or one-locus mismatch unrelated volunteer donors may be an alternative in some patients who lack HLA-matched sib donors. Despite increasing numbers of volunteer unrelated donors in national and international registries, identification of suitable unrelated donors who are matched with the recipient at all HLA-A, -B, -C and -DRB1 loci (8/8 HLA match) or mismatched at one of those loci (7/8 HLA match) is still challenging, especially for patients who are African-American or multiracial. Additionally, the 3- to 4-month delay between initiation of unrelated donor search to HCT is unacceptably long in patients with aggressive hematologic malignancies that are likely to relapse or progress during that interval. Transplantation of single or dual unrelated umbilical cord blood cells (UCB) units is another alternative, although problems with inadequate cell doses, delayed engraftment, graft rejection and infection persist in adult recipients of unrelated UCB transplants.

This is a phase II single-arm open-label study to evaluate the efficacy and safety of haploidentical related allogeneic PBSCT using a nonmyeloablative preparative regimen of intravenous busulfan (Busulfex®), intravenous melphalan (Alkeran®) and intravenous alemtuzumab (Campath®) in subjects who are candidates for related or unrelated allogeneic hematopoietic cell transplantation (HCT; transplantation of bone marrow or PBSCs) but who lack histocompatible related or unrelated donors. This study will also evaluate immunological reconstitution following haploidentical PBSCT by measurement of circulating T cell receptor excision circle (TREC)-positive cells, an indicator of thymic output. Systematic analyses of TREC-positive cells have not been performed in recipients of haploidentical PBSCT after the preparative regimen described in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 75 years.
* one of these diagnoses: acute myeloid leukemia in remission or relapse, acute lymphocytic leukemia in remission or relapse, chronic myeloid leukemia, chronic lymphocytic leukemia, Hodgkin's disease or non-Hodgkin's lymphoma, multiple myeloma, myelodysplastic syndrome, severe aplastic anemia, or paroxysmal nocturnal hemoglobinuria.
* Subjects with hematologic malignancies must have received at least one previous course of chemotherapy or biological therapy (i.e., a subject cannot be enrolled on this study for initial treatment of the malignancy).
* Absence of a healthy related or unrelated volunteer allogeneic donor with whom the subject is either completely HLA matched at HLA-A, -B, -C and -DRB1 (8/8 HLA match) or mismatched at no more than one HLA locus (7/8 HLA match).
* Availability of a healthy haploidentical relative (parent, sib or child) who is able to donate peripheral blood stem cells by apheresis.

Exclusion Criteria:

* Eligibility for another clinical therapeutic protocol or standard-of-care treatment that offers higher probability of cure or long-term control of subject's malignancy.
* Availability of a related or unrelated 7/8 or 8/8 HLA-matched allogeneic donor.
* Severe organ dysfunction
* Untreated or progressive central nervous system involvement by malignancy.
* Subject is pregnant or breast feeding.
* Karnofsky score below 50.
* Seropositivity for human immunodeficiency virus (HIV).
* Life expectancy less than 12 weeks with conventional treatments.
* For subjects who are fertile, refusal to practice contraception upon entering this study and for at least 12 months after PBSCT or after cessation of post-transplant immunosuppressive treatments, whichever occurs later.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2013-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the presence of donor lymphohematopoietic chimerism (defined as at least 50% donor cells in the peripheral blood)in peripheral blood by day +100. | by day +100 (i.e., 100 days after haploidentical PBSCT).

SECONDARY OUTCOMES:
To determine the safety of haploidentical related allogeneic PBSCT using a preparative regimen of busulfan, melphalan and alemtuzumab. | non-relapse mortality at day +100

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Yeager, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center/University Medical Center, Tucson, Arizona, United States